CLINICAL TRIAL: NCT01205958
Title: Clinical Trial to Evaluate the Effect of East-West Collaborative Medicine on Chronic Cervical Pain: a Pilot Study
Brief Title: The Effect of East-West Collaborative Medicine on Chronic Cervical Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Jun-Hwan Lee / Department of Oriental Rehabilitation Medicine, College of Oriental Medicine, Kyung Hee University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KHU 20091458
Record Dates: First submitted 2010-09-14; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Neck Pain
Keywords: Cervical pain; Neck pain; western medicine; oriental medicine; acupuncture; needle
MeSH Terms: conditions — Neck Pain | interventions — Acupuncture Therapy; pyranoprofen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- medication(Zaltoprofen) (Active Comparator)
  Interventions: Procedure: acupuncture
- Acupuncture (Active Comparator)
  Interventions: Procedure: acupuncture
- Zalprofen plus Acupuncture (Active Comparator)
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — Over an three-week period, one group(n=15) gets western medicine treatment(drug medication); another group(n=15) gets oriental medicine treatment(individualized needling 2-3 times a week); the other group(n=15) gets western medicine plus oriental medicine treatment for 3 weeks
  Other Names: Zaltoprofen

SUMMARY:
The purpose of this study is to assess the effect of East-West collaborative medicine on chronic cervical pain.

DETAILED DESCRIPTION:
Design: This is a randomized, controlled study.

Participants: 45 participants with chronic cervical pain are recruited and randomly assigned to three groups.

Intervention: Over an three-week period, one group(n=15) gets western medicine treatment(drug medication); another group(n=15) gets oriental medicine treatment(individualized needling 2-3 times a week); the other group(n=15) gets western medicine plus oriental medicine treatment for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

- presence of Chronic neck pain

Exclusion Criteria:

* Cancer
* Spinal infection
* ankylosing spondylosis
* myelopathy
* moderate hypertension or more
* serious mental disease
* other skeletomuscular disease
* history of operation or acupuncture treatment about spinal disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analogue Scale(VAS) | 7 week

SECONDARY OUTCOMES:
Neck disability index | 7 week
  Neck disability index : questionnaire for measuring how much neck pain affects ability of daily activities
Beck depression inventory | 7 week
  Beck depression inventory : for assessing depression
SF-36 | 7 week
  questionnaire for measuring health-related quality of life
EQ-5D(EuroQol-5 dimension) | 7 week
  questionnaire for measuring health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hwan Lee, OMD, PhD, Principal Investigator — Department of Oriental Rehabilitation Medicine/College of Oriental Medicine/Kyung Hee University
Locations (1):
- Kyunghee University East West Neo Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho JH, Nam DH, Kim KT, Lee JH. Acupuncture with non-steroidal anti-inflammatory drugs (NSAIDs) versus acupuncture or NSAIDs alone for the treatment of chronic neck pain: an assessor-blinded randomised controlled pilot study. Acupunct Med. 2014 Feb;32(1):17-23. doi: 10.1136/acupmed-2013-010410. Epub 2013 Oct 30. PMID 24171895